CLINICAL TRIAL: NCT02812914
Title: NACER II: Reducing Prenatal Exposures to Household Air Pollution in Rural Guatemala Through a Gas Stove/Behavior Intervention to Improve Neonatal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Universidad del Valle, Guatemala (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-17003
Record Dates: First submitted 2016-06-03; First posted 2016-06-24 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Premature Birth; Fetal Growth Retardation; Infections, Respiratory; Exposure to Environmental Pollution, Non-occupational; Infant, Small for Gestational Age
MeSH Terms: conditions — Premature Birth; Fetal Growth Retardation; Respiratory Tract Infections

ARMS (2):
- Phase 1 (Experimental): In Phase I, 25 pregnant women will receive a low-cost gas stove and will be taught by peer educators in group classes how to safely use gas stoves and how to reduce exposure to air pollution.
  Interventions: Other: Low-cost gas stove; Behavioral: Peer education classes
- Phase 2 (Experimental): In Phase 2, the investigators will assess a more resource-intensive behavioral intervention approach with a different group of 25 women who will follow the same study procedures described in Phase I.
  Interventions: Other: Low-cost gas stove; Behavioral: Resource-intensive behavioral intervention approach

INTERVENTIONS:
Other: Low-cost gas stove — Women will be provided with a 3-burner liquid propane gas stove and one year's supply of gas
Behavioral: Peer education classes — Women will participate in four classes on how to safely use gas stoves and methods to reduce exposure to air pollution
  Arms: Phase 1
Behavioral: Resource-intensive behavioral intervention approach — Women will participate in four classes on how to safely use gas stoves and methods to reduce exposure to air pollution. Additionally, peer educators will visit each home after group classes to help the woman, and key decision-makers in her family, identify top priority strategies to reduce air pollution. Using a checklist, peer educators will observe whether household members are adhering to tailored strategies at subsequent home visits, and provide ongoing support to women and their families.
  Arms: Phase 2

SUMMARY:
Greater efforts are needed to bring affordable, clean stoves and adaptive behavioral strategies to the millions of households worldwide that continue to burn solid cooking fuels using inefficient stoves. Two of the leading causes of infant mortality, preterm birth and pneumonia, are associated with high exposures to household air pollution during pregnancy and early infancy. The proposed study will assess the feasibility and acceptability of an introduced liquid petroleum gas stove, complemented by two alternative approaches to delivering tailored behavioral change interventions, among pregnant women and their neonates.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman less than 20 weeks gestation
* Does not smoke cigarettes
* Uses an open fire or deteriorated woodstove for cooking
* Purchases wood
* Intends to stay in the study area for at least one year
* Uses Ministry of Health clinics for routine prenatal care
* Has a mobile phone
* Primary person responsible for cooking in the household
* Able to give Informed Consent

Exclusion Criteria:

* Multiple pregnancy (eg twins)
* Identified as a high-risk pregnancy by physician
* Regularly taking prescription medication
* Smokes cigarettes
* Routinely carries a child less than 2 years old on their back

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04; Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Change in urinary polycyclic aromatic hydrocarbon (PAH) and volatile organic compound (VOC) metabolite concentrations | 1) <20 weeks gestation; 2) 28-32 weeks gestation
Change in 48-hour mean personal carbon monoxide exposure | 1) <20 weeks gestation; 2) 28-32 weeks gestation; 3) Following participation in each behavior change intervention class at 18-24 weeks, 22-28 weeks, and 26-32 weeks gestation; 4) Neonatal after 48 hours, 2 & 4 weeks of life
Change in 48-hour mean kitchen particulate matter concentration | 1) <20 weeks gestation; 2) 28-32 weeks gestation; 3) Following participation in each behavior change intervention class at 18-24 weeks, 22-28 weeks, and 26-32 weeks gestation; 4) Neonatal after 48 hours, 2 & 4 weeks of life
Change in 48-hour mean personal particulate matter exposure | 1) <20 weeks gestation; 2) 28-32 weeks gestation; 3) Following participation in each behavior change intervention class at 18-24 weeks, 22-28 weeks, and 26-32 weeks gestation; 4) Neonatal after 48 hours, 2 & 4 weeks of life
Change in weekly use of gas stoves (cooking events and total cooking time) using temperature loggers | Every month from recruitment to neonatal one month of life (up to 9 months)

SECONDARY OUTCOMES:
Preterm birth | At time of birth (within 48 hours)
Low birth weight | At time of birth (within 48 hours)
Respiratory illness | up to one month following birth

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Thompson, RN, PhD, FNP, Principal Investigator — University of California, San Francisco
Locations (1):
- San Lorenzo Health Center, San Lorenzo, Guatemala

REFERENCES:
- [Derived] Weinstein JR, Diaz-Artiga A, Benowitz N, Thompson LM. Reductions in urinary metabolites of exposure to household air pollution in pregnant, rural Guatemalan women provided liquefied petroleum gas stoves. J Expo Sci Environ Epidemiol. 2020 Mar;30(2):362-373. doi: 10.1038/s41370-019-0163-0. Epub 2019 Sep 2. PMID 31477781
- [Derived] Thompson LM, Diaz-Artiga A, Weinstein JR, Handley MA. Designing a behavioral intervention using the COM-B model and the theoretical domains framework to promote gas stove use in rural Guatemala: a formative research study. BMC Public Health. 2018 Feb 14;18(1):253. doi: 10.1186/s12889-018-5138-x. PMID 29444650